CLINICAL TRIAL: NCT02310971
Title: A Phase 2 Trial of Cvac (Autologous Dendritic Cells Pulsed With Recombinant Human Fusion Protein [Mucin 1-Glutathione S-Transferase] Coupled to Oxidized Polymannose) in Patients With Resected Stage I or Stage II Adenocarcinoma (Cancer) of the Pancreas
Brief Title: Cvac as Maintenance Treatment Patients With Resected Stage I or Stage II Adenocarcinoma (Cancer) of the Pancreas
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial has been terminated per Sponsor direction due to longer than expected clinical and regulatory approvals.
Sponsor: Prima BioMed Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAN-301
Record Dates: First submitted 2014-11-15; First posted 2014-12-08 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Pancreatic Carcinoma Stage I; Pancreatic Carcinoma Stage II
Keywords: Adenocarcinoma, resected
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Biologic/Vaccine (Experimental): Cvac will be administered via intradermal injection, every 4 weeks for the first 3 doses and thereafter every 12 weeks for 3 additional doses for a total of 6
  Interventions: Biological: CVac

INTERVENTIONS:
Biological: CVac — Cvac will be administered via intradermal injection, every 4 weeks for the first 3 doses and thereafter every 12 weeks for 3 additional doses for a total of 6

SUMMARY:
The purpose of this study is to assess the safety and tolerability of CVac, an investigational cell therapy, in patients with resected stage I or II adenocarcinoma of the pancreas who have completed surgery with or without front-line chemotherapy or radiation therapy.

After confirmation of non-measurable disease patients will undergo leukapheresis for manufacture of the study agent.

DETAILED DESCRIPTION:
A total of approximately 40 patients at up to 30 clinical sites will be screened for eligibility into the study within 6 weeks of completing treatment, including R0 (complete resection with no microscopic residual tumor) or R1 (complete resection with no grossly visible tumor but microscopically positive margins) surgery for stage I or stage II adenocarcinoma of the pancreas with or without chemotherapy and radiation. Eligible patients must have no measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (Eisenhauer 2009) and tumor marker carbohydrate antigen 19-9 [CA 19-9] not greater than 2 × the upper limit of normal (ULN) following surgery with or without chemotherapy or radiation. Prior surgery, neoadjuvant chemotherapy, adjuvant chemotherapy, and radiation therapy are allowed.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically diagnosed adenocarcinoma of the pancreas, stage I or stage II disease
2. Postoperative confirmed R0 or R1 resection status with no evidence of residual disease based on radiographic Imaging
3. CA 19-9 less than 2 × the ULN by the central laboratory
4. No greater than 6 weeks since completion of prior therapy, which includes surgery with or without radiation or chemotherapy
5. Mucin 1-positive tumor as determined by central immunohistopathology. Sites will be asked to submit archival tissue (patients may start the study if tissue is available at an outside hospital, but not yet requested or received)
6. Signed an informed consent form (ICF)
7. Willing and able to complete study procedures within the study timelines
8. Life expectancy of at least 6 months in the investigator's opinion
9. ≥ 18 years of Age
10. ECOG performance status < 2 (Karnofsky ≥ 70%)
11. Normal organ and marrow function: serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × ULN and serum bilirubin ≤ 1.5 × ULN unless Gilbert's syndrome has previously been confirmed for the patient, white blood cells (WBCs) ≥ 3.0 K/µL, absolute neutrophil count (ANC) ≥ 1.0 × 109/L, hemoglobin ≥ 8 g/dL, and platelets ≥ 100 × 109/L
12. Not pregnant, and if of childbearing potential, agrees to use a highly effective method of birth control (implanted, injectable, or oral combination hormonal method alone or in possible combinations, intrauterine device, vasectomized partner, or abstinence) prior to study entry, for the duration of the study, and for 3 months after the last dose of Cvac. Male partners of a study patient must use a condom in addition to the acceptable method of contraception for the female partner as specified above

Exclusion Criteria:

1. Active, acute, or chronic clinically significant infections or bleeding
2. Uncontrolled hypertension (systolic blood pressure > 150 mmHg or diastolic blood pressure > 100 mmHg) or history of congestive heart failure (≥ Grade 2)
3. Active angina pectoris, stroke, or recent myocardial infarction (within 6 months)
4. Additional uncontrolled, serious medical or psychiatric illness
5. Evidence or history of central nervous system metastases
6. Inadequate renal function defined as a creatinine clearance < 60 mL/min as determined by the central laboratory
7. Additional malignancy diagnosed within 5 years of study enrollment, except carcinoma in situ of the cervix or basal cell and squamous cell carcinomas of the skin
8. Treatment with any other investigational agent (for any condition) within 4 weeks of Screening
9. Infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV), or syphilis (Treponema pallidum [TPHA])
10. Concurrent systemic treatment with steroids or other immunosuppressant agents at a dose considered by the investigator to be higher than a standard physiological dose
11. Active autoimmune disease; any previous autoimmune disease must not require chronic treatment in the 6 months prior to screening
12. Germany only:

Oversensitivity to the substances or another component of the investigational medicinal product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Assessment of safety and tolerability of CVac. (adverse events, vital signs, 12 lead ECG, relevant changes in physical examination) | 10-12 months
  Safety analyses will be performed on the Safety Population. Safety and tolerability will be summarized using descriptive statistics and or listed and assessed by adverse events, vital signs, 12 lead ECG, relevant changes in physical examination.

SECONDARY OUTCOMES:
Assessment of Progression-Free Survival (PFS) and Overall Survival (OS) following the initiation of Cvac in this patient population | Participants will be followed from baseline until death from any cause or end of study, whichever comes first, assessed approximately every 12 weeks for up to 36 month
  The efficacy endpoints for this pilot study include OS and PFS, PFS is defined as the time from baseline to the date of radiological scan used to determine Progressive disease evaluated approximately every 12 weeks after baseline.

OTHER OUTCOMES:
Evaluation of the time to next treatment (TTNT) | Baseline until end of Progression free survival for up to 36 months
Evaluation of the immunologic response to Cvac administration in this patient population | Baseline until end of Progression free survival for up to 36 months
  Descriptive statistics will be used to summarize the changes in immunologic Response.
Investigation of biomarkers, including tumor and immune characteristics, of clinical efficacy of Cvac in this patient population | Baseline until end of Progression free survival for up to 36 months
  Immunologic parameters will be evaluated as exploratory efficacy endpoints. Plasma, serum, and tissue (i.e., tumor sample collected during surgery) samples will be collected and will be used for immunological assays.
Assessment of the change in quality of life (QoL) following the initiation of Cvac in this patient population | Baseline until end of Progression free survival for up to 36 months
  Quality-of-life scores will be calculated based on the QLQ-C30 and Module QLQ-PAN26 scoring manuals. The QoL scores will be summarized. descriptively. Data permitting, the QoL scores may be evaluated longitudinally using a linear mixed-effects model for repeated measurements.